CLINICAL TRIAL: NCT01140503
Title: An Open Label Study Evaluating the Safety and Efficacy of Apremilast in the Treatment of Cutaneous Disease in Patients With Dermatomyositis
Brief Title: A Study to Evaluate the Safety and Efficacy of Apremilast in the Treatment of Skin Disease in Patients With Dermatomyositis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment of participants
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Fiorentino, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-03302010-5522; 16975
Record Dates: First submitted 2010-04-06; First posted 2010-06-09 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- apremilast (Experimental): apremilast 20mg bid
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast 20mg PO BID

SUMMARY:
This study is designed to evaluate the safety and efficacy of an oral medicine (called apremilast) for treating skin involvement in patients with the disease dermatomyositis.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Must be 18 years at time of signing informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* Patients must have a diagnosis of DM based upon the characteristic cutaneous findings proposed by Sontheimer1 and a skin biopsy consistent with DM
* Subjects must be a candidate for systemic therapy for their DM skin disease: a subject is considered a candidate, if, in the judgment of the investigator, they are not adequately responding to aggressive sun protection along with the use of potent (e.g. class I or II) topical corticosteroids and/or immunomodulators
* Must have cutaneous disease activity of at least "moderate" on a 5 point Likert scale (using the PGA)
* Must have cutaneous disease activity score of at least 5 on the CDASI (activity) scale
* Concurrent therapy with topical corticosteroids and/or prednisone and/or antimalarials is permitted as defined in Exclusion Criteria.
* Concurrent therapy with methotrexate azathioprine, mycophenolate mofetil, or leflunomide is permitted as defined in Exclusion Criteria
* Must meet the following laboratory criteria:

  * Hemoglobin ≥ 12 g/dL
  * White blood cell (WBC) count ≥ 3000 /uL (≥ 3.0 X 10^9/L) and < 14,000/uL (< 14 X 10^9/L)
  * Platelets ≥ 100,000 /uL (≥ 100 X 10^9/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Total bilirubin ≤ 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]) ; 1.5x upper limit of normal (ULN) unless, in the opinion, of the investigator, the elevation is secondary to active muscle inflammation.
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner. A FCBP must agree to have pregnancy tests every 28 days while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication

Exclusion Criteria:

* History of inadequate response of cutaneous DM disease to greater than 2 of the following agents: methotrexate, cyclosporine, azathioprine, mycophenolate mofetil, IVIG, leflunomide, cyclophosphamide.
* History of inadequate response to thalidomide for dermatomyositis skin disease.
* Receiving topical therapy within 14 days of Study Day 0 (including but not limited to topical corticosteroids, tacrolimus, pimecrolimus). Exceptions: low potency corticosteroids will be allowed as background therapy for treatment of the face and scalp as needed, but dose must be stable 14 days prior to Study Day 0 and throughout the study
* Concurrent therapy with prednisone (or equivalent dose of systemic corticosteroid) at greater than 10 mg daily.
* Concurrent therapy with more than one of the following agents: methotrexate, azathioprine, mycophenolate mofetil, leflunomide.
* Receiving the following dosages of medications during the study or within 28 days before Study Day 0:

  * Hydroxychloroquine at >600 mg/day
  * Chloroquine at >400 mg/day
  * Methotrexate at >25 mg/week
  * Mycophenolate mofetil at >3 g/day
  * Azathioprine at >3 mg/kg/day
  * Leflunomide at >20mg/day
* Treatment with the following biologic agents:

  * Adalimumab, etanercept, efalizumab, or infliximab within 12 weeks of Study Day 0 and for the study duration
  * IVIG within 12 weeks of Study Day 0 and for the study duration
  * Rituximab within 9 months of Study Day 0 and for the study duration
  * Alefacept within 24 weeks of Study Day 0 and for the study duration
* Have received fluctuating doses of any of the following medications 28 days before Study Day 0: methotrexate, mycophenolate mofetil, azathioprine, leflunomide, dapsone
* Have received fluctuating doses of hydroxychloroquine 2 months before Study Day 0
* Have received fluctuating doses of chloroquine 3 months before Study Day 0
* Have received fluctuating doses of prednisone within 14 days prior to Study Day 0
* Received leflunomide >20 mg/day in the 6 months prior to Study Day 0
* Treatment with any investigational drug therapy within 28 days before Study Day 0 or biologic therapies within 30 days or 5 half-lives of the biologic agent, whichever is longer, before Study Day 0
* Currently receiving any of the following medications:

  * Cyclophosphamide
  * Intravenous immunoglobulin (IVIG)
  * Any TNF inhibitor, including adalimumab, etanercept, infliximab, or certolizumab
  * Rituximab
  * Efalizumab
  * Cyclosporine
  * Oral FK506 (tacrolimus)
  * Thalidomide
* History of any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major uncontrolled disease
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding
* Latent Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative (PPD) skin test.
* History of active Mycobacterium tuberculosis infection (any subspecies) within 3 years prior to the screening visit and without documentation of successful treatment

  * Subjects who completed treatment at least 3 years prior to screening but lack documentation may not be enrolled in the study. Subjects who completed treatment at least 3 years prior to screening are allowed if successful treatment was completed at least 3 years prior to screening and is documented and available for verification
* History of incompletely treated latent Mycobacterium tuberculosis infection as indicated by:

  * Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis
  * Subject's self reported history of incomplete treatment for Mycobacterium tuberculosis
* Any clinically significant abnormality on 12-lead ECG at screening
* Presence of hepatitis B surface antigens (HBsAg) or Hepatitis B core antibody positive at screening
* Antibodies to hepatitis C virus at screening
* History of human immunodeficiency virus (HIV) infection
* Malignancy or history of malignancy except for treated (i.e. cured) basal-cell skin carcinomas
* Abnormal chest x-ray findings other than that consistent with dermatomyositis-associated interstitial lung disease. Chest x-rays performed within 3 months prior to start of study drug are acceptable
* Any condition, including the presence of laboratory abnormalities, that places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Franklin Fiorentino, Principal Investigator — Stanford University; Katharine Arefiev, Sub-Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single center study in which patients were recruited from a clinical practice. Participant recruitment lasted from December, 2009 until August, 2011. The first patient was screened in February, 2010 and the last patient visit was in July, 2011.
Groups:
- Apremilast: All subjects received apremilast 20mg PO BID
Period: Overall Study
Arm/Group | Apremilast
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Physician Global Assessment of Skin Activity (VAS) [Median (Standard Deviation); unit: units on a scale] — This is a visual analog scale (0-10cm) in which the physician estimates the global activity of the dermatomyositis skin disease. The score ranges from 0 to 10, with higher scores representing higher disease severity
  units on a scale | 3.8 (0.98)
Physician Global Assessment of Skin Activity (Likert) [Median (Standard Deviation); unit: units on a scale] — This is a 5 point scale (0=clear; 1=mild; 2=moderate; 3=severe; 4=very severe) in which the physician estimates the severity of the dermatomyositis skin disease activity
  units on a scale | 2 (0)
CDASI Activity Score [Median (Standard Deviation); unit: units on a scale] — This is a validated instrument (Cutaneous Dermatomyositis Activity and Severity Index) quantifying dermatomyositis skin disease activity by assigning severity points on redness, scale, and ulceration to specific body sites typically involved by dermatomyositis. Possible scores for the CDASI-a range from 0 to 100, with higher numbers represent higher severity of skin disease. Scores above 15 are considered to have moderate-to-severe activity. A clinically meaningful improvement in this scale is 4.
  units on a scale | 31 (6.8)
Manual Muscle Testing (MMT-8) score [Median (Standard Deviation); unit: units on a scale] — This is a validated measure of muscle strength. Scale goes from 0-150. 150 is perfect strength.
  units on a scale | 147 (4.21)
Patient Pruritis Scale (VAS) [Median (Standard Deviation); unit: units on a scale] — This is a patient-reported estimate of itching. The patient fills out a visual analog scale (0-10cm) to estimate the severity of itching. A higher score is more severe itch.
  units on a scale | 2.9 (2.40)
Dermatology Life Quality Index (DLQI) [Median (Standard Deviation); unit: units on a scale] — This is a validated instrument that estimates the impact of skin disease on the quality of life. score ranges from 0-30, with a higher score representing a greater adverse impact on quality of life.
  units on a scale | 9 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Analysis Will be Safety, as Measured by the Number of Adverse Events and Serious Adverse Events Occuring During 12 Weeks of Therapy and 4 Weeks of Followup.
Time Frame: 16 weeks
Measure: Number; unit: adverse events
Arm/Group | Apremilast
Number analyzed (Participants) | 5
adverse events | 12

2. Secondary Outcome: The Secondary Outcome Measure Will be Efficacy, as Measured by the Number of Participants Experiencing a 30% Decreased in the CDASI-a Score at 12 Weeks.
Description: This was an intent to treat analysis--dropouts are considered treatment failures. Missing data at 12 weeks imputed by last observation carried forward.
Time Frame: Data collected at 12 weeks after baseline visit.
Measure: Number; unit: participants
Arm/Group | Apremilast
Number analyzed (Participants) | 5
participants | 1

3. Secondary Outcome: The Secondary Outcome Measure Will be Efficacy as Measured by the Mean Change in CDASI-activity at 12 Weeks
Description: The CDASI (Cutaneous Dermatomyositis Activity and Severity Index) is a validated instrument to measure skin disease activity in dermatomyositis. A clinically meaningful change is a decrease of 4 points. All missing data are imputed using last observation carried forward. Calculation is performed as the score at 12 weeks minus the score at baseline.
Time Frame: Data collected at baseline at 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 5
units on a scale | 6 (4)

ADVERSE EVENTS:
Arm/Group | Apremilast
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=5)
headache (Nervous system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine headache (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Left Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1 (1)
Elevated serum creatinine (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to low enrollment. Therefore we only have data on 5 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less